CLINICAL TRIAL: NCT06268652
Title: Patient Derived Organoid-guided Personalized Treatment Versus Treatment of Physician's Choice in Patients With Relapsed and Refractory Breast Cancer：a Multicenter, Randomized, Controlled Phase III Trial
Brief Title: Patient Derived Organoid-guided Personalized Treatment Versus Treatment of Physician's Choice in Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Yanxia, Principal Investigator, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B2023-686-01
Record Dates: First submitted 2024-01-23; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Refractory Breast Carcinoma
Keywords: breast cancer; TPC; patient derived organoid; PDO
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Capecitabine; Vinorelbine; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organoid-guided personalized treatment (Experimental): Subjects randomly assigned to OGPT need to provide sufficient tissue for organoid culture. After successful organoid culture, drug screening will be performed, and they will be treated with drugs predicted to be sensitive by PDO drug susceptibility screening.
  Interventions: Other: Organoid-guided personalized treatment
- Treatment of physician's choice (Active Comparator): Subjects in the TPC arm will receive treatment with one of the following regimens selected by the physician following NCCN guidelines: capecitabine, gemcitabine, vinorelbine, and eribulin. If it is HER2-positive, anti-HER2 therapy can be combined with it, except for ADC drugs.
  Interventions: Drug: Gemcitabine; Drug: Capecitabine; Drug: Vinorelbine; Drug: Eribulin

INTERVENTIONS:
Other: Organoid-guided personalized treatment — After the organoid culture is successful, the personalized drug library customized by our team will be used for screening. Sensitive drugs are selected based on the results of drug screening, and the most appropriate personalized treatment plan is selected based on NCCN guideline recommendations, drug safety, and conventional drugs used in the treatment of breast cancer. The personalized drug library customized by our team contains 55 drugs approved by the FDA. For specific usage, dosage and time intervals, please refer to the instructions of the corresponding drug.
  Other Names: OGPT
  Arms: Organoid-guided personalized treatment
Drug: Gemcitabine — 1000mg/m2，IV, days 1, 8, q3w
  Other Names: Gemzar
  Arms: Treatment of physician's choice
Drug: Capecitabine — 1000mg/m² , PO, bid, days1-14, q3w
  Other Names: Xeloda
  Arms: Treatment of physician's choice
Drug: Vinorelbine — 25mg/m2, IV or 60mg/m² (oral), days 1 and 8, q3w
  Other Names: Navelbine
  Arms: Treatment of physician's choice
Drug: Eribulin — 1.4mg/m², IV, days 1 and 8, q3w
  Other Names: Halaven
  Arms: Treatment of physician's choice

SUMMARY:
This multicenter, open-label, randomized phase III trial is designed to study the efficacy and safety of organoid-guided personalized treatment （OGPT）versus treatment of physician's choice (TPC) in previously treated refractory breast cancer.

DETAILED DESCRIPTION:
This multicenter, open-label, randomized phase III trial is designed to study the efficacy and safety of organoid-guided personalized treatment （OGPT）versus treatment of physician's choice (TPC) in previously treated refractory breast cancer. Molecular subtype, presence of visceral metastases, and number of prior chemotherapy treatments for advanced or metastatic disease will stratify randomization. subjects in the OGPT arm will receive the treatment predicted to be the most effective by PDO drug sensitivity screening, and subjects in the TPC arm will receive treatment of physician's choice. The primary population to be included in the study will be patients with refractory breast cancer who have received multiple lines of prior therapy and who have at least one measurable target lesion according to RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent form
2. Aged over 18 years old, regardless of gender;
3. Locally advanced or metastatic breast cancer confirmed by histopathology;
4. Received ≥2 previous lines of anti-tumor treatment and developed resistance to standard treatment;
5. Life expectancy ≥3 months;
6. ECOG performance status 0 to 2;
7. Have measurable or/and evaluable lesions (non-radiotherapy target areas) (lesion evaluation is based on Recist1.1 standards);
8. No serious organ (main organ: heart, lung, liver, kidney) functional abnormalities (refer to respective standards);
9. Routine blood test: white blood cells (WBC) ≥3 × 109/L; absolute neutrophil count (ANC) ≥1.5 × 109/L; platelets (PLT) ≥100 × 109/L; hemoglobin (Hgb) ≥8g /dL;
10. Blood biochemical indicators: AST (SGOT), ALT (SGPT) ≤ 2.5 × upper limit of normal value (ULN) (in the case of no liver invasion) or ≤ 5 × upper limit of normal value (ULN) (in the case of liver invasion) Bottom); total bilirubin (TBIL) ≤ ULN; serum creatinine clearance calculated according to the CG formula > 30 mL/min
11. Coagulation function: prothrombin time (PT), international normalized ratio (INR) ≤ 1.5 × ULN (unless warfarin is being used for anticoagulation);
12. Able to comply with the research visit plan and other program requirements;
13. All patients of childbearing age must agree to take effective contraceptive measures during the study and within 6 months of stopping treatment. Female patients of childbearing age must have a negative urine pregnancy test before treatment.

Subjects must meet all of the following additional criteria to be included in the OGPT group:

1. No absolute contraindications to tissue-invasive procedures required to obtain organoid cultures。
2. Sufficient tissue can be provided for organoid culture: biopsy samples (length >1cm, 3 strips), surgical resection samples (total volume >1cm3, weight >0.2g), thoracentesis, abdominal puncture, pericardiocentesis and other malignant effusion samples (pleural effusion >500mL, ascites >500m) and confirmed to contain malignant tumor cells.

Exclusion Criteria:

1. The medical history and comorbidities are as follows:

   1. The patient is participating in other interventional clinical studies or the end of treatment in the previous clinical study is less than 4 weeks;（2）Those who have been treated less than 4 weeks since the last anti-tumor treatment (radiotherapy, chemotherapy, targeted therapy, immunotherapy or local-regional treatment); the adverse reactions related to anti-tumor treatment (except alopecia) after previous systemic anti-tumor treatment have not returned to NCI- Patients with CTC AE ≤ grade 1;
   2. Other active malignant tumors that require simultaneous treatment;
   3. Known history of organ transplantation and allogeneic hematopoietic stem cell transplantation;
   4. For subjects who have undergone major surgery or severe trauma, the effects of the surgery or trauma have been eliminated for less than 14 days before enrollment;
   5. Patients with active pulmonary tuberculosis need to be excluded. Patients suspected of having active pulmonary tuberculosis should have chest X-rays, sputum, and clinical symptoms and signs to rule out the disease. Patients with a history of active pulmonary tuberculosis infection within the previous year must be excluded, even if they have been treated; patients with a history of active pulmonary tuberculosis infection more than 1 year ago must also be excluded, unless it is proven that the course and type of anti-tuberculosis treatment previously used are satisfactory. appropriate;
   6. Severe acute or chronic infection requiring systemic treatment
   7. Suffering from heart failure (New York Heart Association Class III or IV) and despite receiving appropriate medical treatment, poorly controlled coronary artery disease or arrhythmia, or a history of myocardial infarction within 6 months before screening patient.
2. Pregnant or lactating women.
3. No anti-tumor treatment is planned.
4. Known to have a positive history of human immunodeficiency virus (HIV) test or known to have acquired immunodeficiency syndrome (AIDS);
5. Untreated active hepatitis (hepatitis B: HBsAg positive and HBV DNA ≥ 500IU/mL; hepatitis C: HCV RNA positive and abnormal liver function); combined with hepatitis B and hepatitis C co-infection;
6. Hypersensitivity to any study drug;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Within approximately 48 months
  Progression-free survival (PFS) is defined as the time from the date of the first dose to the earlier of the dates of the first objective documentation of radiographic progressive disease (PD) or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Within approximately 48 months
  Overall survival (OS) is defined as the time from the date of first dose to the date of death from any cause.
Objective Response Rate (ORR) | Within approximately 48 months
  The number of participants with objective response is assessed every six weeks from Cycle 1 Day 1 through discontinuation of treatment. Objective response rate (ORR) was defined as the proportion of participants who achieved a best overall response of complete response or partial response based on local radiologists/investigators' tumor assessments.
Duration of Response (DOR) | Within approximately 48 months
  Duration of response was defined as the time interval between the date of first documentation of objective response (CR or PR) and the date of the first objective documentation of disease progression or death due to any cause.
Disease Control Rate (DCR) | Within approximately 48 months
  Disease Control Rate (DCR) was defined as the percentage of patients who have achieved complete response, partial response and stable disease
Incidence of Treatment-related Adverse Events | Within approximately 48 months
  Incidence of Treatment-related Adverse Events as assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Shi, Principal Investigator — Sun Yat-sen University
Locations (1):
- Yanxia Shi, Guangzhou, None Selected, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT06268652/Prot_000.pdf
  • Informed Consent Form (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT06268652/ICF_001.pdf